CLINICAL TRIAL: NCT02929550
Title: Predicted Impact on Cardiovascular and Economic Outcomes of Swedish Atherosclerotic Cardiovascular Disease Guideline 2014 With Focus on Lipid Lowering Treatment
Brief Title: Impact of Guidelines on Cardiovascular and Economic Outcomes With Focus on Lipid Lowering Drugs
Acronym: GuLLD
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Gunilla Journath, Postdoc, Karolinska Institutet
Other Study IDs: 2015/4:7
Record Dates: First submitted 2016-10-07; First posted 2016-10-11 (Estimated); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Acute Myocardial Infarction
Keywords: Cardiovascular disease; Costs; Guidelines; Lipids; Myocardial infarction
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction | interventions — Non-Randomized Controlled Trials as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Well-controlled cohort (LDL-C ≤ 1.8 mmol/L): Individuals in the Swedish Secondary Prevention after Heart intensive care Admission (SEPHIA) is a sub register within SWEDEHEART collecting data on secondary prevention and cardiac rehabilitation with well-controlled LDL-cholesterol
  Interventions: Other: Well-controlled
- Non-controlled cohort: Individuals in the Swedish Secondary Prevention after Heart intensive care Admission (SEPHIA) is a sub register within SWEDEHEART collecting data on secondary prevention and cardiac rehabilitation and with not well-controlled LDL-C

INTERVENTIONS:
Other: Well-controlled — Both groups got treatment but well-controlled reached target of LDL-C<1.8 mmol/l
  Other Names: Non-controlled
  Groups: Well-controlled cohort (LDL-C ≤ 1.8 mmol/L)

SUMMARY:
Methods: All patients <75 years registered in the Swedish Secondary Prevention after Heart Intensive care Admission registry (SEPHIA), will be followed-up within one year post-myocardia infarction (MI). The REACH risk prediction and a calibrated model for recurrent cardiovascular disease (CVD) events and death will be used to estimate base case, and calibrated CVD outcomes based on gender-specific risk factors. The predicted impact of the LDL-C reduction on the risk of CVD will be based on Cholesterol Treatment Trialists´ Collaboration findings.

DETAILED DESCRIPTION:
SWEDEHEART is a Swedish national registry consisting of several sub registries in which patients with acute coronary syndrome are prospectively registered. Patient characteristics, hospital treatments, drug treatments at discharge, and outcome for patients consecutively included and treated at all Swedish coronary care units are collected in this registry.SEPHIA is a sub registry collecting data on secondary prevention and cardiac rehabilitation. Follow-up are registered at six to ten weeks and at 12 to14 months post MI by office visits or phone. Around 80 % of all Swedish acute myocardial infarction (AMI) patients below the age of 75 years are included in this register.

In this study, a cohort of 5 904 (74% men) registered in the SEPHIA registry and who had one year follow-up during 2013, will be included. Data are aggregated and delivered from the SWEDEHEART/SEPHIA national registry. All patients were informed about their participation in the registry, the follow-up, and their right to decline participation. No written consent was obtained

ELIGIBILITY:
Inclusion Criteria: All patients with acute myocardial infarction registered in the SEPHIA registry and who had one year follow-up during 2013 -

Exclusion Criteria:none

-

Max Age: 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: a cohort of 5 904 (74% men) registered in the Swedish Secondary Prevention after Heart Intensive Care Admission (SEPHIA) registry and who have had one year follow-up during 2013
Sampling Method: Non-Probability Sample
Enrollment: 5304 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Percentage of AMI patients who have achieved target goal of LDL-cholesterol 1.8 mmol/L or not | AMI patients with one year follow-up year 2013
  Treatment gap will be analysed in well-controlled (LDL-C ≤1.8 mmol/L) and non-controlled ( LDL-C >1.8 mmol/L) cohort in men and women separately.

SECONDARY OUTCOMES:
Number of predicted CVD events gained if target LDL-cholesterol was achieved in the non-controlled group | Predicted number of events within a 10 year period
  Number of events predicted to occur in the non-controlled group
Health care costs in SEK saved, due to number of predicted CVD events gained if target LDL-cholesterol was achieved in the non-controlled group | Predicted health care costs within a 10 year period
  Health care costs predicted to be gained if the non-controlled group achieved target LDL-cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Gunilla Journath, PhD, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Journath G, Hambraeus K, Hagstrom E, Pettersson B, Lothgren M. Predicted impact of lipid lowering therapy on cardiovascular and economic outcomes of Swedish atherosclerotic cardiovascular disease guideline. BMC Cardiovasc Disord. 2017 Aug 16;17(1):224. doi: 10.1186/s12872-017-0659-2. PMID 28814290
- See also: Predicted impact of lipid lowering therapy on cardiovascular and economic outcomes of Swedish atherosclerotic cardiovascular disease guideline. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5559790/pdf/12872_2017_Article_659.pdf